CLINICAL TRIAL: NCT00485966
Title: A Phase 2, Multi-Center, Open Label Study Evaluating Clinical Efficacy, Safety, and Pharmacodynamic Effects of Quarfloxacin (CX-3543) in Patients With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Study Evaluating Effects of CX-3543 in Patients With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn prior to patient enrollment
Sponsor: Cylene Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3-07-001
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: Adult Leukemia; CLL; B-CLL; Chronic Lymphocytic Leukemia; B-cell CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, B-Cell | interventions — CX 3543

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CX-3543 — 360 mg/m2 daily x 5 q 21 days

SUMMARY:
This is a Phase 2, open-label, multicenter, efficacy, safety, and pharmacodynamic study of CX-3543 in patients with relapsed or refractory B-cell chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the response rate, safety, pharmacodynamic effects, and duration of response of CX-3543 in patients with relapsed or refractory B-cell CLL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell CLL with indications for treatment by National Cancer Institute (NCI) Working Group criteria.
* Measurable disease (lymphocytes ≥ 5,000/microliter, or palpable lymphadenopathy or bone marrow involvement > 30%).
* Males and females 18 years of age or older.
* Received a minimum of one prior purine analog-based chemotherapy regimen (e.g., fludarabine, cladribine, or pentostatin) and one monoclonal antibody therapy (e.g., Campath or Rituxan) but ≤ 4 chemotherapy regimens.
* Patients must have central intravenous (IV) access, or agree to the insertion of a central line.
* All previous cancer therapies, radiation, hormonal therapy and surgery, must have been discontinued at least 28 days prior to the start of treatment. Any cytotoxic chemotherapy must have been discontinued 28 days prior to the start of treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1 above baseline.
* Normal oxygen saturation with pulse oximetry on room air.
* Hemoglobin ≥ 9 gm/dL (may be post-transfusion).
* Platelet count ≥ 25,000/microliter.
* Total bilirubin < 2 X upper limit of normal (ULN), and ALT and AST < 2 x ULN.
* Serum creatinine within normal limits OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above the upper normal limit for the institution
* ECOG Performance Status ≤ 1.
* Anticipated survival of at least 3 months.
* For men and women of child-producing potential, use of effective contraceptive methods during the study and for one month after discontinuation of treatment.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return to the clinic for required assessments.

Exclusion Criteria:

* Pregnant or nursing women.
* Severe chronic obstructive pulmonary disease with hypoxemia or an uncorrectable pulmonary compromise.
* Seizures not controlled by anticonvulsant therapy.
* Participation in any investigational drug study within 28 days before quarfloxacin administration.
* Patients with second malignancy requiring active treatment.
* Active symptomatic bacterial, fungal, or viral infection including active HIV or viral (A, B, or C) hepatitis.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis.
* Patients who have exhibited allergic reactions to a similar structural compound (e.g., fluoroquinolones) or formulation (containing buffers and/or polyethylene glycol).
* Patients with life- or function-threatening CLL complications (e.g., cord compression, hemolytic crisis, urinary tract obstruction).
* Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any of the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy
Safety

SECONDARY OUTCOMES:
Clinical benefit
Pharmacodynamics
Study drug blood levels
Progression free survival

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Oregon Health and Sciences University, Portland, Oregon
  - Cancer Therapy and Research Center, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin